CLINICAL TRIAL: NCT06813313
Title: Randomized Controlled Trial of Two Accelerated Transcranial Magnetic Stimulation Methods in the Treatment of Resistant Depression: Intermittent Theta Burst Stimulation With an 8-Coil Versus H1-Coil
Brief Title: Theta Burst Stimulation With an 8-Coil Versus H1-Coil for Resistant Depression
Acronym: rTBShTBS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dominique JANUEL (Other)
Responsible Party: Sponsor-Investigator, Dominique JANUEL, Head of clinical research department, Centre hospitalier de Ville-Evrard, France
Organization: Centre hospitalier de Ville-Evrard, France (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-A00954-43
Record Dates: First submitted 2025-01-27; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Treatment of Resistant Depression; H1-Coil; Theta Burst Stimulation
Keywords: Resistant Depression; H1-Coil; Theta burst stimulation; TMS; Accelerated Transcranial Magnetic Stimulation; Intermittent Theta Burst Stimulation with an 8-Coil versus H1-Coil
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS ARM (Other): The treatment consists of 8 sessions per day for 5 days, with daily self-assessments for 1 week. Each session lasts approximately 9 minutes and 50 seconds with a 50-minute break between sessions. The application of rTBS will be done using the Cool-B65 coil, targeting the DLPFC region identified by neuronavigation.
  Interventions: Device: repetitive transcranial magnetic stimulation
- hTBS Arm (Other): The treatment consists of 8 sessions per day for 5 days, with daily self-assessments for 1 week. Each session lasts approximately 9 minutes and 50 seconds with a 50-minute break between sessions. The application of hTBS will be done using the H1 coil, targeting the DLPFC region located 6 cm forward from the motor cortex.
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — A burst of 3 pulses sent at a frequency of 50 Hz, repeated with a frequency of 5 Hz for 2 seconds, followed by an 8-second pause. This sequence is repeated for 59 cycles, totaling 9 minutes and 50 seconds, with a total of 1800 pulses.

SUMMARY:
The goal of this clinical trial is to compare response rates after treatment with Figure Eight-Coil TMS versus H-Coil TMS on the prefrontal cortex left dorsolateral, in patients suffering from depression resistant. The main question it aims to answer is:

rTBS (accelerated neuronavigated intermittent Theta Burst Stimulation) is more effective than hTBS (accelerated deep intermittent Theta Burst Stimulation) in the treatment of resistant depression in terms of response rate.?

Researchers will compare Figure Eight-Coil TMS (rTBS) versus H-Coil TMS (hTBS) to see if rTBS is more effective than hTBS.

Participants will:

* Receive, for each stimulation method, 8 sessions per day spaced 50 minutes apart, over 5 days.
* Have visit all day of stimulation for checkups and tests.
* Have a a research MRI before and after treatment.
* Have follow-up visits at 1 month, 2 months, 3 months, 6 months, and 12 months post-treatment, via teleconsultation.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Presenting a major depressive episode according to the DSM-5-TR criteria, occurring as part of major depressive disorder (unipolar depression)
* The major depressive episode must meet the criteria for treatment resistance, defined by a lack of response to at least two different antidepressant treatments prescribed at an effective dose for a duration of 6 weeks or more
* Stable treatment for at least 6 weeks
* Affiliation with a social security system or State Medical Assistance (Aide Médicale d'État)
* Patient agrees to participate in the study and has signed an informed consent form

Exclusion Criteria:

* Presence of a contraindication to TMS: epilepsy, intracranial foreign body, cochlear implant, retinal implant, pacemaker
* Presence of a bipolar disorder according to DSM-5-TR criteria
* Presence of catatonic or psychotic features during the current episode
* Presence of severe psychiatric disorders other than a major depressive episode
* Presence of neurological disorders
* Unstable epilepsy
* Current moderate to severe addiction disorders other than caffeine and/or tobacco
* Current suicidal ideation
* Use of any brain stimulation treatment (ECT, rTMS, tDCS) for the current episode
* Pregnancy or breastfeeding
* Women of childbearing potential without effective contraception
* Persons under guardianship or legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-02-16 (Estimated); Primary Completion 2027-11-18 (Estimated); Study Completion 2028-11-18 (Estimated)

PRIMARY OUTCOMES:
The response rate according to the MADRS scale | Before the treatment and after the treatment at 5 day.
  The response rate is defined as an improvement of more than 50% compared to baseline on the MADRS clinical scale (Montgomery-Asberg Depression Rating Scale). The MADRS consists of 10 items, each scored from 0 to 6 : depressive mood, appetite, sleep, psychomotor retardation, anxiety, suicidal thoughts, cognitive impairment, pessimism, loss of control and demoralization. The total score is the sum of the scores for all 10 items. The overall score can range from 0 to 60.
  0 to 6: No depression 7 to 19: Mild depression 20 to 34: Moderate depression 35 to 60: Severe depression

SECONDARY OUTCOMES:
Clinical improvement of treatment-resistant depression | Before the treatment and after the treatment at 5 days.
  We use:
  - MADRS (Montgomery-Åsberg Depression Rating Scale) : Remission: A MADRS score of less than 10.
Clinical improvement of treatment-resistant depression | Before the treatment and after the treatment at 5 days.
  We use:
  - HDRS-17 (Hamilton Depression Rating Scale - 17 items): The scale contains 17 items, each scored on a scale from 0 to 4, 0 to 2, or 0 to 3, depending on the item. The total score is obtained by adding the scores of all 17 items. The total score can range from 0 to 52.
  Response: A reduction of 50% or more in the total HDRS-17 score compared to baseline is generally considered a response to treatment.
  Remission: A score of 7 or less is typically considered remission from depression.
Clinical improvement of treatment-resistant depression | Before the treatment and after the treatment at 5 days.
  We use:
  - QIDS-SR : The patient answers the 16 items, each assessing various depressive symptoms, and the score ranges from 0 to 27, based on their experiences over the past week. A 50% reduction in the total score from baseline is considered a response.
Clinical improvement of treatment-resistant depression | Before the treatment and after the treatment at 5 days.
  We use:
  - EQ5D : The EQ-5D is a brief tool for assessing health-related quality of life. It measures 5 key dimensions of health.
Tolerance to treatment | Each visits of clinical trial : each day of treatment (5 days), at 1 month, 2 month, 3 month, 6 month and 12 month.
  Rate of adverse effects and rate of premature withdrawal from the study.
Improvement of cognitive functions. | Before the treatment and after the treatment at 5 day.
  Trail Making Test A and B (version from the Group for the Evaluation of Executive Functions, GREFEX, Army individual test 1944, based on Godefroy, 2012)
Improvement of cognitive functions. | Before the treatment and after the treatment at 5 day.
  Free Recall / Cued Recall at 16 items (RL/RI-16), version A or B
Improvement of cognitive functions. | Before the treatment and after the treatment at 5 day.
  Stroop Test (Golden, 1978)
Improvement of cognitive functions. | Before the treatment and after the treatment at 5 day.
  Wisconsin Card Sorting Test (WCST), GREFEX version
Improvement of cognitive functions. | Before the treatment and after the treatment at 5 day.
  N-back Task (version from the Attention Assessment Tests, TAP)
Improvement of cognitive functions. | Before the treatment and after the treatment at 5 day.
  Go/No-Go Inhibition Task (TAP version)
Improvement of cognitive functions. | Before the treatment and after the treatment at 5 day.
  Digit Span and "Coding" subtest from the Wechsler Adult Intelligence Scale (WAIS-IV)
Improvement of cognitive functions. | Before the treatment and after the treatment at 5 day.
  Verbal Fluency Test (GREFEX version)
Improvement of neurophysiological functions | Before the treatment and after the treatment at 5 day.
  Variation in brain functional connectivity between baseline and the end of the rTMS treatment.
Improvement of neurophysiological functions | Before the treatment and after the treatment at 5 day.
  Neurobiological/neurophysiological variables: change in heart rate variability.
Improvement of neurophysiological functions | Before the treatment and after the treatment at 5 day.
  Change in serum BDNF levels.
Improvement of neurophysiological functions | Before the treatment and after the treatment at 5 day.
  Change in motor cortex neuroexcitability.
Pain detection and pain tolerance using an experimental pain task | Before the treatment and after the treatment at 5 day.
  Cold pain using the cold pressor task and mechanical pain using the algomete